CLINICAL TRIAL: NCT03117205
Title: The Effect of Kinesio Taping® on Motor Control in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Claudio Cazarini Junior, Principal Investigator, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36422114.2.0000.5512
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2014-09

CONDITIONS: Knee Injuries; Pain Syndrome
MeSH Terms: conditions — Knee Injuries; Somatoform Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping® group (Experimental)
  Interventions: Other: Application of Kinesio Taping®
- placebo group (Placebo Comparator)
  Interventions: Other: Kinesio Taping® placebo application

INTERVENTIONS:
Other: Application of Kinesio Taping® — The technique was applied following the methods described in the original method for patellofemoral instability
  Arms: Kinesio Taping® group
Other: Kinesio Taping® placebo application — Simulation of the application of the Kinesio Taping® technique.
  Arms: placebo group

SUMMARY:
Background: Recently, several professionals are using the Kinesio Taping® in the treatment of pathologies related to the knee, aiming to improve the motor control, increase the response of muscle activation and promoting better joint stability.

Purpose: The objective of this study is to evaluate the effect of the application of Kinesio Taping® in motor control of patients with patellofemoral pain syndrome.

Methods: This is a 2-arm, randomized with a blinded assessor. We selected 40 women with patellofemoral pain (age 25.2±4,years) were randomly assigned to one of two groups: placebo group (n= 20) and the Kinesio Taping® group (n=20). The placebo group received the application of a non-stretchable tape (Micropore) crosswise on the thigh and the Kinesio Taping® group followed all the criteria of the method in placing the bandage. All patients received the evaluation of the motor control banding pre and post a patch, by means of the method Y balance test.

ELIGIBILITY:
Inclusion Criteria:

* Patellofemoral pain syndrome diagnoses
* Aged 18-40 years
* Kujala questionnaire above

Exclusion Criteria:

* Neurological disorders
* BMI indicating obesity (BMI> 30kg / m²)
* High-performance athletes
* History of surgeries in lower limbs
* In treatment of any underlying pathology

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Method Y balance test | Evaluation was performed after 30 minutes of applying the bandage
  Was used the method of evaluating motor control known as Y test